CLINICAL TRIAL: NCT03734328
Title: Platelet Rich Fibrin Accelerates Wound Healing and Reduces Postoperative Complications of Palatal Subepithelial Connective Tissue Donor Site: a Controlled Randomized Clinical Trial
Brief Title: Evaluation of the Effects of Platelet Rich Fibrin on the Palatal Mucosal Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, AYSAN LEKTEMUR ALPAN, Assistant Proffessor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 60116787-020/44407
Record Dates: First submitted 2018-11-03; First posted 2018-11-07 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Wound Healing; Pain, Postoperative; Bleeding Wound
Keywords: connective tissue graft; platelet rich fibrin; patient perceptions; VAS
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- connective tissue graft (Active Comparator): Drug:local anesthesia (2% lidocaine with 1:100,000 epinephrine/ultracaine ds ampule)
  Other names:
  * 5/0 silk suture
  Interventions: Procedure: connective tissue graft; Procedure: connective tissue graft&PRF; Other: connective tissue graft&PRF
- connective tissue graft&PRF (Experimental): Drug: local anesthesia (2% lidocaine with 1:100,000 epinephrine/ultracaine ds ampule)
  Other names:
  -5/0 silk suture
  Interventions: Procedure: connective tissue graft; Procedure: connective tissue graft&PRF; Other: connective tissue graft&PRF

INTERVENTIONS:
Procedure: connective tissue graft — * anesthesia of the palatal mucosa
  * subepithelial connective tissue graft harvesting
  * suturing (5/0 silk suture)
Procedure: connective tissue graft&PRF — anesthesia of the palatal mucosa subepithelial connective tissue graft harvesting
  -suturing (5/0 silk suture)
Other: connective tissue graft&PRF — * taking blood from patient
  * centrifuging blood
  * obtain PRF

SUMMARY:
Subepithelial connective tissue graft (SCTG) has greater predictability for root coverage and causes minimal discomfort to patient. Although donor site heals with primary intention causing less scar tissue, in some different harvesting procedures primary flap closure may not be achieved due to nature of thick palatal tissues. Some potential complications may occur at donor site such as: necrosis of graft and palatal site, pain, excessive hemorrhage, protracted discomfort, donor site infection and in some cases donor site paresthesia. Platelet rich fibrin (PRF) is a platelet concentrate obtained by a simple procedure that does not require biochemical blood involvement.Based on the known biological effects of PRF, the aim of this study is to evaluate the PRF in the management of soft tissue donor sites in term of bleeding and pain sensation, and to observe the changes in tissue healing after a subepithelial connective tissue graft procedure at palatal donor site.

DETAILED DESCRIPTION:
Successful treatment of gingival recession (GR) is based on the use of clinically predictable periodontal plastic surgery (PPS) procedures. There are many procedures and different surgical procedures were proposed. Coronally advanced flap and subepithelial connective tissue graft (SCTG) is a good combination to increase the keratinized tissue width and reduce the amount of gingival recession.

SCTG has greater predictability for root coverage and causes minimal discomfort to patient. Although donor site heals with primary intention causing less scar tissue, in some different harvesting procedures primary flap closure may not be achieved due to nature of thick palatal tissues.

Some potential complications may occur at donor site such as: necrosis of graft and palatal site, pain, excessive hemorrhage, protracted discomfort, donor site infection and in some cases donor site paresthesia.

Platelet rich fibrin (PRF) is a platelet concentrate obtained by a simple procedure that does not require biochemical blood involvement. The three-dimensional fibrin network and presence of many growth factors such as fibroblast growth factor, platelet-derived growth factor (PDGF) and epidermal growth factor supports effective neovascularization, accelerated wound closure and rapid cicatricial tissue remodeling. The strong fibrin architecture distinguishes it from other kinds of platelets concentrates and it seems responsible for the slow release of growth factors over a period of 7-14 days5. This period is seen as sufficient to prevent complications after connective tissue graft. Since the first description by Choukroun in 2000, PRF has been used in the clinical field for more than a decade in oral surgery and implant dentistry.

Based on the known biological effects of PRF, the aim of this study is to evaluate the PRF in the management of soft tissue donor sites in term of bleeding and pain sensation, and to observe the changes in tissue healing after connective tissue graft procedure at palatal donor site.

ELIGIBILITY:
Inclusion Criteria:

* who needed connective tissue graft for treating gingival recessions were included

Exclusion Criteria:

* Patients with systemic disorders (immunologic diseases, uncontrolled diabetes mellitus, ongoing chemotherapy or radiotherapy),
* smoking,
* nausea
* pregnancy/lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Defining wound healing to 40 patient with early healing index | 14 days
  to inspect the early wound healing on donor site on palate using early healing index on 3rd, 7th and 14th postoperatively. (1) complete flap closure, no fibrin line in the interproximal area; (2) complete flap closure, fine fibrin line in the interproximal area; (3) complete flap closure, fibrin clot in the interproximal area; (4) incomplete flap closure, partial necrosis of the interproximal tissue; and (5) incomplete flap closure, complete necrosis of the interproximal tissue
postoperative pain | 10 days
  Patients were instructed to complete pain diary for the day at the surgery, first day, third day, seventh day, tenth day after surgery. The visual analog scale (VAS) that consists of a 10-cm line anchored by 2 extremes was used for perception measurements . Total score was 100 and less score was 0 according to this scale. According to this scale "0" means no pain, no discomfort during chewing and speaking, while the "100",meant 'worst pain, extreme discomfort during chewing and speaking'

SECONDARY OUTCOMES:
postoperative bleeding | 7days
  Patients were told to record DB, 'present' or 'absent' in a 7-day postoperative period.

OTHER OUTCOMES:
Tissue colour match | 14 days
  On days 3, 7, 14 , the color of the palatal mucosa was assessed by the VAS score with the adjacent and opposite mucosa color. In this evaluation, 0 points showed no color matching, and 100 points showed excellent color matching with evaluated tissues

CONTACTS AND LOCATIONS:
Overall Officials: Murat AKGUL, prof. dr., Principal Investigator — Pamukkale University Faculty of Dentistry Department of Periodontolgy
Locations (1):
- Pamukkale University Faculty of Dentistry, Denizli, Deni̇zli̇, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choukroun J, Diss A, Simonpieri A, Girard MO, Schoeffler C, Dohan SL, Dohan AJ, Mouhyi J, Dohan DM. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part IV: clinical effects on tissue healing. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e56-60. doi: 10.1016/j.tripleo.2005.07.011. PMID 16504852
- [Background] Femminella B, Iaconi MC, Di Tullio M, Romano L, Sinjari B, D'Arcangelo C, De Ninis P, Paolantonio M. Clinical Comparison of Platelet-Rich Fibrin and a Gelatin Sponge in the Management of Palatal Wounds After Epithelialized Free Gingival Graft Harvest: A Randomized Clinical Trial. J Periodontol. 2016 Feb;87(2):103-13. doi: 10.1902/jop.2015.150198. Epub 2015 Aug 27. PMID 26313017